CLINICAL TRIAL: NCT02317211
Title: Effect of Purified Anthocyanin on Oxidative Stress and Glycemic Control in Subjects With Type 2 Diabetes Mellitus: A Randomized, Double-Blinded, Placebo-Controlled Trial
Brief Title: Purified Anthocyanins Supplementation in Type 2 Diabetes Mellitus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shaoguan University (Other)
Responsible Party: Principal Investigator, Di Li, PhD, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZXYZM-1
Record Dates: First submitted 2014-12-07; First posted 2014-12-15 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus，Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): placebo 320 mg daily for twelve weeks
  Interventions: Dietary Supplement: placebo
- anthocyanins treatment (Experimental): anthocyanin supplement 320mg daily for twelve weeks
  Interventions: Dietary Supplement: Anthocyanin

INTERVENTIONS:
Dietary Supplement: Anthocyanin — Extract of blueberry and huckleberry （MEDOX，http://www.medox.no/english）
  Other Names: natural purified anthocyanin
  Arms: anthocyanins treatment
Dietary Supplement: placebo — starch
  Other Names: placebo capsule
  Arms: control

SUMMARY:
Anthocyanins, the water-soluble compounds that make plants appear different colors, have been shown to prevent insulin resistance, reduce the blood glucose and oxidative stress in rodents. The purpose of our study is to evaluate a potential protective effect of purified anthocyanins supplement on type 2 diabetes mellitus patients.

DETAILED DESCRIPTION:
The study was designed as a randomized, double-blind label, interventional study on patients with T2DM. The eligible Participants are randomly assigned to control and Anthocyanins supplement group. During the 12 weeks trial period,the participants were instructed to consume two anthocyanin capsules or placebo capsules twice daily (30 min after breakfast and supper).

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with type 2 diabetes mellitus according to the Chinese type 2 diabetes prevention guide 2010, diagnostic criteria are as follows:(1) Diabetes symptoms (polydipsia, polyphagia, polyuria, weight loss, skin itching, blurred vision and other acute metabolic network disorder that caused by high blood sugar)combined with random blood sugar ≥11.1 OR,(2)fasting plasma glucose(FPG)≥7.0 OR (3)2h blood sugar after oral glucose tolerance test(OGTT)≥ 11.1
* Subject is between 25 and 75 years of age, inclusive.
* Subject BMI is ≥18.5 kg/m2 and ≤35 kg/m2

Exclusion Criteria:

* Subject that is diagnosed as type 1 diabetes, gestational diabetes and other kinds of diabetes expect type 2.
* Subject that use exogenous insulin for glucose control.
* Subject that has a history of diabetic ketoacidosis.
* Subject that has coronary artery disease, mental disorder, cancer, cirrhosis, renal disease and hepatic disease.
* Subject that has had operation less than six months prior to screening visit.
* Subject that uses supplementation with vitamins or antioxidants.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Glycemic Control | Twelve weeks
  Hemoglobin A1c (HbA1c),fasting blood glucose (FBG) at study entry and 12 weeks after dietary intervention

SECONDARY OUTCOMES:
Biomakers related to oxidative stress | Twelve weeks
  Superoxide dismutase (SOD),Glutathione peroxidase (GSH-PX)
Blood lipids | Twelve weeks
  Cholesterol, HDL-cholesterol, Triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Di Li, PhD, Principal Investigator — Guangdong Provincial Key Laboratory of Food, Nutrition and Health; Department of Nutrition, School of Public Health, Sun Yat-Sen University (Northern Campus)

REFERENCES:
- [Derived] Li D, Zhang Y, Liu Y, Sun R, Xia M. Purified anthocyanin supplementation reduces dyslipidemia, enhances antioxidant capacity, and prevents insulin resistance in diabetic patients. J Nutr. 2015 Apr;145(4):742-8. doi: 10.3945/jn.114.205674. Epub 2015 Feb 4. PMID 25833778